CLINICAL TRIAL: NCT05258058
Title: Mitigating Cancer-Related Cognitive Impairment in Older Adults With Cancer: Memory and Attention Adaptation Training-Geriatrics (MAAT-G) Phase I
Brief Title: Feasibility of the Memory and Attention Adaptation-Training Geriatrics Intervention in Older Cancer Survivors With Mild Cognitive Impairment
Acronym: urochester
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allison Magnuson (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor-Investigator, Allison Magnuson, Associate Professor - Department of Medicine , Hematology/Oncology (SMD), University of Rochester
Organization: University of Rochester (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UCCS19102- Part 2; K76AG064394-03S1 (NIH)
Record Dates: First submitted 2022-02-17; First posted 2022-02-28 (Actual); Results first posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-06

CONDITIONS: Cognitive Dysfunction
Keywords: cancer-related cognitive difficulties; mild cognitive impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MAAT-G Intervention (Experimental): MAAT-G Workshops & participant workbook use (8 workshops)
  Interventions: Behavioral: Memory and Adaptation Training-Geriatrics

INTERVENTIONS:
Behavioral: Memory and Adaptation Training-Geriatrics — MAAT-G is a cognitive behavioral therapy-based intervention comprised of 10 workshop sessions as well as a participant workbook. The workshop sessions are delivered one on one by a health professional via videoconferencing technology.
  Other Names: MAAT-G

SUMMARY:
Cancer-related cognitive dysfunction (CRCD) affects up to 75% of patients receiving chemotherapy and older adults are at greater risk of developing CRCD, which can negatively affect their functional independence and quality of life. Memory and Attention Adaptation Training-Geriatrics (MAAT-G) is a cognitive behavioral therapy-based intervention tailored specifically for older adults and the feasibility of MAAT-G in older cancer survivors with Mild Cognitive Impairment (MCI) is being evaluated.

DETAILED DESCRIPTION:
Cancer-related cognitive dysfunction (CRCD) affects up to 75% of patients receiving chemotherapy and older adults are at greater risk of developing CRCD, which can negatively affect their functional independence and quality of life. Memory and Attention Adaptation Training-Geriatrics (MAAT-G) is a cognitive behavioral therapy-based intervention tailored specifically for older adults. MAAT-G is a series of 10 workshops delivered by a trained health profession via videoconferencing technology. The feasibility of MAAT-G in older cancer survivors with Mild Cognitive Impairment (MCI) is being evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Be age 65 or older
2. Able to provide informed consent. All patients will be assessed using the University of California, San Diego Brief Assessment of Capacity to Consent (UBACC)56 - a score >14.5 will define ability to independently provide informed consent. For patients scoring <14.5, or if investigators have additional concerns, we will require that their health care proxy participate in the consenting process and sign an informed consent and patients will required to provide assent.
3. Able to read and understand English
4. Have a prior diagnosis of cancer and completed curative intent chemotherapy. Patients are permitted to be receiving maintenance therapy (e.g. endocrine therapy) in the adjuvant setting.
5. Have a clinical diagnosis of MCI, a score <26 on the Montreal Cognitive Assessment (MOCA), or a score <18 on the Montreal Cognitive Assessment-BLIND (MOCA-BLIND). If the patient had a MOCA evaluation completed as a part of routine clinical care in the preceding 3 months prior to consent date, this may be used for eligibility purposes.
6. Be independent in Activities of Daily Living (ADL)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-12-10 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allison Magnuson, Principal Investigator — Univ. of Rochester Wilmot Cancer Center
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Groups:
- MAAT-G Intervention: MAAT-G Workshops & participant workbook use (10 workshops)
  Memory and Adaptation Training-Geriatrics: MAAT-G is a cognitive behavioral therapy-based intervention comprised of 10 workshop sessions as well as a participant workbook. The workshop sessions are delivered one on one by a health professional via videoconferencing technology.
Period: Overall Study
Arm/Group | MAAT-G Intervention
Started | 12
Completed | 10
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | MAAT-G Intervention
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.8 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: MAAT-G Feasibility Completion Rate
Description: Evaluate the feasibility of MAAT-G in older cancer survivors with mild cognitive impairment by determining study completion rate of this population.
Time Frame: 10 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | MAAT-G Intervention
Number analyzed (Participants) | 12
Participants | 10

2. Secondary Outcome: Proportion of Patients Who Described at Least One MAAT-G Skill
Description: To obtain descriptive feedback on the usability of the intervention and guide further adaptation, qualitative interviews with patients and their caregivers (if available) will be conducted at completion of the intervention.
Time Frame: 10 Weeks
Population: Two patients withdrew from the study and therefore not included in the population.
Measure: Count of Participants; unit: Participants
Arm/Group | MAAT-G Intervention
Number analyzed (Participants) | 10
Participants | 9

3. Secondary Outcome: Change in Cognitive Function (Pre-Post Changes Functional Assessment of Cancer Therapy-Cognition [FACT-Cog])
Description: Examine the pre-post change in perceived and objective cognitive function in older cancer survivors with MCI using the Functional Assessment of Cancer Therapy-Cognition (FACT-Cog version 2): a 37 item scale assessing perceived cognitive impairment (Total score range 0-185, higher score indicates better cognitive function). Mean change from baseline score is reported.
Time Frame: 10 Weeks
Population: Two patients withdrew from the study and therefore not included in the population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MAAT-G Intervention
Number analyzed (Participants) | 10
score on a scale | 6.39 (12.20)

4. Secondary Outcome: Mean Usability
Description: Enhance our understanding of the usability of a telehealth CRCD intervention (including barriers and facilitators) for older cancer survivors with MCI and the perceived MAAT-G intervention effect using the System Usability Scale (SUS) (a score on a 10-item scale, with a total score ranging from 0-100; a higher score corresponds to greater usability).
Time Frame: 10 Weeks
Population: Two patients withdrew from the study and therefore not included in the population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MAAT-G Intervention
Number analyzed (Participants) | 10
score on a scale | 78.75 (15.332)

5. Primary Outcome: MAAT-G Intervention Adherence Rate
Description: Evaluate the feasibility of MAAT-G in older cancer survivors with mild cognitive impairment by determining the study intervention adherence rate of this population (proportion of MAAT-G workshops completed).
Time Frame: 10 Weeks
Measure: Number; unit: percentage of workshops adhered to
Units Other Than Participants: workshops
Arm/Group | MAAT-G Intervention
Number analyzed (Participants) | 12
Number analyzed (workshops) | 120
percentage of workshops adhered to | 88.33

ADVERSE EVENTS:
Time Frame: 10 weeks
Arm/Group | MAAT-G Intervention
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-03-15): https://cdn.clinicaltrials.gov/large-docs/58/NCT05258058/Prot_SAP_000.pdf
  • Informed Consent Form (2023-03-20): https://cdn.clinicaltrials.gov/large-docs/58/NCT05258058/ICF_001.pdf